CLINICAL TRIAL: NCT01166620
Title: Observational Real-world Evaluation of Cost of Infections of RA Patients on Biologics
Brief Title: Observational Real-world Evaluation of Cost of Infections of Rheumatoid Arthritis (RA) Patients on Biologics
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-244
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients with rheumatoid arthritis new to abatacept.
- Patients with rheumatoid arthritis new to etanercept
- Patients with rheumatoid arthritis new to adalimumab
- Patients with rheumatoid arthritis new to infliximab

SUMMARY:
To quantify the incremental cost of infections in patients treated with etanercept, adalimumab or infliximab versus abatacept.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older;
* Have a diagnosis of of rheumatoid arthritis (ICD-9:714x.xx);
* Have been enrolled for at least 6 months for the 6 months assessment and 12 months for the 12 months assessment;
* are enrolled in a health plan between February 2006 and June 2009
* have claims indicating at least one use of either abatacept, etanercept, adalimumab or infliximab for at least 6 months for teh 6 months assessment and 12 months for the 12 months assessment

Exclusion Criteria:

* Patients not continuously eligible for health plan benefits for the same evaluation periods will be excluded
* Patients who are on other biologics in the 6 and 12 month post-index period will be excluded (ex. those in the abatacept cohort will be excluded if they also have claims for etanercept in the 6 and 12 month post-index period).
* Patients on biologics 6 months prior to the biologic index date will also be excluded
* Patients with diagnosis for other non-RA conditions commonly treated with biologics (ex. Crohn's disease) during the 6 month pre-index period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial health plan members
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incremental total and component (inpatient, outpatient and pharmacy) direct costs due to infection in patients treated with etanercept, adalimumab or infliximab versus abatacept | 6 months
Incremental total and component (inpatient, outpatient and pharmacy) direct costs due to infection in patients treated with etanercept, adalimumab or infliximab versus abatacept. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm